CLINICAL TRIAL: NCT00378586
Title: Barrier Function and Production of Inflammatory Cytokines in the Rectal Mucosa in Patients With Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Michael Ibsen, Rigshospitalet
Other Study IDs: KA-05037
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Rectal biopsy — Rectal biopsy.
Procedure: Measurement of inflammatory markers in the rectal mucosa — IL-6, TNF-alfa.
Procedure: Measurement of rectal lactic acid — Equilibrium dialysis.

SUMMARY:
Life-threatening infection impairs bloodflow to the gut, thereby causing less delivery of oxygen. This leads to increased formation of different inflammatory and infectious markers.

The investigators hypothesize, therefore, that there is a significant difference in the concentrations of inflammatory and infectious markers in the rectal mucosa between patients with septic shock and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock

Exclusion Criteria:

* Age < 18 years
* No next of kin
* Pathology of the descending or sigmoid colon or rectum
* Pregnancy
* 1st degree relatives with inflammatory bowel disease
* Severe coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Septic shock patients.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ibsen, MD, Principal Investigator — Dept. of Intensive Care 4131, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Dept. of Intensive Care 4131, Copenhagen, Denmark